CLINICAL TRIAL: NCT07182318
Title: Validation and Application of the FIGO Nutrition Checklist in the Third Trimester Pregnant Women.
Brief Title: Validation of the FIGO Nutrition Checklist in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Katarzyna Skorupska, MD PhD, Medical University of Lublin
Other Study IDs: 01/2025
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; Nutrition
Keywords: pregnancy; nutrition; child health; maternal health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- third trimester pregnant women: ither outpatients attending the obstetrics clinic or inpatients at the Department of Obstetrics and Gynecology at the Independent Public Health Care Facility in Puławy.
  Interventions: Diagnostic Test: The FIGO Nutrition Checklist
- At the time of dietary assessment, the mean gestational age was 35 weeks ± 3 days
  Interventions: Diagnostic Test: The FIGO Nutrition Checklist

INTERVENTIONS:
Diagnostic Test: The FIGO Nutrition Checklist — patient fulfilled the questionnaire twice. period of time 2-3 days
  Other Names: The FIGO Nutrition Checklist after 2-3 days

SUMMARY:
The aims of this study were to verify the test-retest reproducibility of FIGO Nutrition Checklist as well as evaluate dietary habits of pregnant women in the third trimester.

DETAILED DESCRIPTION:
The FIGO Nutrition Checklist was developed to evaluate nutrient intake in both the preconception and gestational periods. It allows to identify inadequate diets as well as provides feedback to women on their dietary habits. The questionnaire is available in several lenguages including polish.

The checklist employs a binary response format-"Yes" or "No." Negative responses may indicate potential nutritional deficits requiring further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* gestational age was 35 weeks ± 3 days.

Exclusion Criteria:

* terminal disease of the baby
* diabetes
* severe hypertension
* IUGR

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: either outpatients attending the obstetrics clinic or inpatients at the Department of Obstetrics and Gynecology at the Independent Public Health Care Facility in Puławy
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
test-retest reproducibility | 2 to 3 days between fulfillment of the questionnaire
  In most questions of the polish version of FIGO Nutrition Checklist the test-retest reproducibility was very good or excellent. Number patients who changed answers between the first and the second asssesment varied from 0 to 12.5%. The minimum-0% and maximum values-100%. The differences were not statistically significant (McNemar's test)

SECONDARY OUTCOMES:
An analysis of dietary habits was conducted using the FIGO Nutrition Checklist. | 2-3 days
  The dietary habits of the pregnant participants were analyzed using the FIGO Nutrition Checklist, with a focus on the consumption of specific food groups. The questionnaire comprises four sections: dietary requirements, anthropometric measurements (including body weight and height), and six questions assessing diet quality. The final section evaluates folic acid supplementation, sunlight exposure, and indicators of anemia among respondents. The checklist uses a binary response format ("Yes" or "No"), where negative responses may indicate potential nutritional deficiencies that warrant further assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michał Bogusiewicz, Professor, Study Director — Medical University of Lublin
Locations (1):
- Samodzielny Publiczny Zakład Opieki Zdrowotnej w Puławach, Puławy, Poland

IPD SHARING:
Plan to Share IPD: Yes
we plan to publish the data
Supporting Information: Study Protocol, CSR
Time Frame: we plan to publish i 2025 year
Access Criteria: everybody who will read the publication

REFERENCES:
- [Background] International Federation of Gynecology and Obstetrics (FIGO). FIGO Nutrition Checklist: A tool for assessing nutrition in women of reproductive age. International Journal of Gynecology & Obstetrics, 2017: 137(2), 218-223